CLINICAL TRIAL: NCT05424042
Title: Health, Aging and Later-Life Outcomes Pilot Trial (HALLO-P): A 9-month Randomized Pilot Trial of 3 Nutritional Interventions in 120 Older Adults With an Indication for Weight Loss
Brief Title: Health, Aging and Later-Life Outcomes
Acronym: HALLO-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB00072563; U01AG073240 (NIH)
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Results first posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Aging
Keywords: older adults; caloric restriction; time restricted eating
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: One-hundred participants (100) will be randomized to the three study arms in a 1:1:1 ratio. Recruitment will be stratified by sex. Once eligibility is established and baseline testing is completed, participants will be randomized using a permuted block scheme with blocks of varying size stratified by sex to one of the 3 intervention groups.
Who Masked: Outcomes Assessor
Masking Description: Staff who will assess outcomes at follow up visits will be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- In-Person Caloric Restriction Arm (Experimental): This group will undergo a 9-month behavioral diet intervention targeting a 20% reduction in caloric intake. During the first 6 months, participants will meet in-person one time each month individually and three times/month in a group setting with a dietitian and/or behavioral coach. During the remaining three months of intervention, there will be one group and one individual meeting each month. Participants will keep diet records using the Fitbit app on a tablet and weight using a BodyTrace™ smart scale that transmits data through a study-specific Companion App. Participants will use wrist-worn Fitbit step monitors to track their physical activity and receive feedback via the app, with a goal to promote movement across the day, continuously increasing their daily step count.
  Interventions: Behavioral: In-Person Caloric Restriction
- Remote Caloric Restriction Arm (Experimental): This group will have a 20% reduction in caloric intake and meeting schedule, and physical activity goal similar to the In-Person group. However, the remote arm intervention will be delivered via video conferencing.
  Interventions: Behavioral: Remote Caloric Restriction
- Time-Restricted Eating Arm (Experimental): This group will undergo a 9-month dietary intervention targeting consumption of all daily caloric intake within an 8-hour window of time, with no restrictions on caloric intake. During the first 6 months, participants will meet in-person once per month individually and three times per month in a group setting with a dietitian and/or behavioral coach. During the remaining 3 months of intervention, there will be one group and one individual meeting each month. Participants in TRE will be asked to log into the study-specific Companion App each day to document the beginning and end of their feeding cycles with timing of meals/snacks consumed. As in the CR arms, participants will use wrist-worn Fitbit step monitors to track their physical activity and receive feedback via the app, with a goal to promote movement across the day, increasing daily step count. Continuous glucose monitoring will be used at intervals to document glucose levels over a 7-10-day period.
  Interventions: Behavioral: Time-restricted

INTERVENTIONS:
Behavioral: In-Person Caloric Restriction — 20% CR delivered in-person by dietitian/coach
  Arms: In-Person Caloric Restriction Arm
Behavioral: Remote Caloric Restriction — 20% reduction in caloric intake, meeting schedule, and physical activity goal delivered remotely.
  Arms: Remote Caloric Restriction Arm
Behavioral: Time-restricted — 8-hour TRE with ad libitum caloric intake. This group will undergo a 9-month dietary intervention targeting consumption of all daily caloric intake within an 8-hour window of time, with no restrictions on caloric intake.
  Arms: Time-Restricted Eating Arm

SUMMARY:
The purpose of this pilot research is to test the feasibility of two interventions focused on either reducing total calorie intake or reducing the total time that calories are ingested each day in older adults. Participation in this research will involve visits to our clinic for testing and weekly intervention visits (in-person or remote depending on group assignment) for nine months with total participation lasting about a year.

DETAILED DESCRIPTION:
This pilot study is part of a larger planning process to design a full-scale randomized trial to evaluate the long-term effects of caloric restriction (CR) and time restricted eating (TRE) on the health of older adults. The specific objective of the HALLO-P is to collect data to inform the design of the full-scale randomized trial to evaluate the long-term effects of caloric restriction and time restricted eating in older adults. The pilot is a 9-month clinical trial. The pilot data will be used to refine recruitment criteria, estimate recruitment yields, and refine intervention approaches.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling men and women residing in Forsyth County, NC or surrounding counties
* obesity (BMI = 30 - < =40 kg/m2) or are overweight (BMI = 27 - <30 kg/m2 with an indication for weight loss (e.g., hypertension, hyperlipidemia, elevated waist girth, controlled diabetes)

Exclusion Criteria:

* persons for whom the interventions are potentially unsafe
* history of eating or nutritional disorders
* those who are likely to drop out due to severe chronic illness or other reasons
* who show inability to perform self-monitoring activities required by the interventions
* those doing shift work because disturbances in circadian cycles may interfere with TRE
* uncontrolled or previously undetected diabetes because disease management may interfere with the interventions
* certain medical treatments may complicate outcome interpretation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B. Kritchevsky, PhD, Principal Investigator — Wake Forest University Health Sciences; Barbara J. Nicklas, PhD, Principal Investigator — Wake Forest University Health Sciences; Michael E. Miller, PhD, Principal Investigator — Wake Forest University Health Sciences; W. Jack Rejeski, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Wake Forest Baptist Hospital, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stowe CL, Kennedy K, Emilson SS, Neiberg RH, Kritchevsky SB, Miller ME, Houston DK, Nicklas BJ, Fanning J, Rejeski WJ; HALLO-P Investigators. The Health, Aging, and Later-Life Outcomes Pilot Study: Design, recruitment, and participants' baseline characteristics. Contemp Clin Trials. 2025 Oct;157:108049. doi: 10.1016/j.cct.2025.108049. Epub 2025 Aug 18. PMID 40834924

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in July 2022 at one clinical site.
Pre-assignment Details: Participants were pre-screened on the phone and then brought in for consent then two screening visits which included a run in period prior to randomization to groups.
Period: Overall Study
Arm/Group | In-Person Caloric Restriction Arm | Remote Caloric Restriction Arm | Time-Restricted Eating Arm
Started | 22 | 34 | 34
Completed | 20 | 34 | 29
Not Completed | 2 | 0 | 5
Not completed — Withdrawal by Subject | 2 | 0 | 4
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | In-Person Caloric Restriction Arm | Remote Caloric Restriction Arm | Time-Restricted Eating Arm | Total
Number analyzed (Participants) | 22 | 34 | 34 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (5.0) | 68.7 (4.6) | 66.1 (5.0) | 67.2 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 21 | 22 | 56
  Male | 9 | 13 | 12 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 5 | 14
  White | 18 | 29 | 28 | 75
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 22 | 34 | 32 | 88
  Unknown or Not Reported | 0 | 0 | 0 | 0
Screening Weight [Mean (Standard Deviation); unit: kg] | 90.5 (11.9) | 90.8 (14.0) | 89.7 (12.7) | 90.3 (4.9)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 31.0 (2.9) | 31.7 (2.9) | 32.0 (2.9) | 31.7 (2.9)
Total MoCA Score [Mean (Standard Deviation); unit: points] — Montreal Cognitive Assessment (MoCA): The MoCA questionnaire is used to exclude any participant with impaired cognition that would preclude them from participating. The MoCA test is a 30-point test administered in approximately 10 minutes which assesses several cognitive domains including short-term memory recall task, visuospatial abilities, executive functions, attention, concentration, and working memory, language, and orientation to time. A score <22 would exclude the participant.
  points | 26.0 (1.9) | 26.2 (2.0) | 26.0 (2.1) | 26.1 (2.0)
Grip Strength [Mean (Standard Deviation); unit: kg] | 32.1 (8.8) | 32.1 (11.3) | 30.3 (7.8) | 31.4 (9.4)
Step Count per day [Mean (Standard Deviation); unit: steps per day] | 7201 (2536) | 6411 (1888) | 7327 (2960) | 6962 (2514)
eSPPB [Mean (Standard Deviation); unit: score] — The expanded Short Physical Performance Battery consists of standing balance tasks (side-by-side, semi- and full-tandem stands), a 4-m walk to assess usual gait speed, and time to complete 5 repeated chair stands. The SPPB was expanded to increase the holding time of the standing balance tasks from 10 to 30 seconds and added a single leg stand and a narrow walk test of balance to minimize ceiling effects of the SPPB. The eSPPB scores are continuous and range from 0 to 4, with higher scores indicative of better performance
  score | 2.58 (0.35) | 2.49 (0.31) | 2.59 (0.36) | 2.55 (0.34)
400 meter Fast Walk Time [Mean (Standard Deviation); unit: seconds] | 292.4 (42.4) | 305.2 (42.2) | 398.7 (36.4) | 299.8 (40.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Sustained >10% Caloric Restriction
Description: Ability of participants to sustain Caloric Restriction >10%
Time Frame: Month 9
Population: The TRE Arm did not participate in caloric restriction and are not included in the outcome analysis. Only those participants with data from baseline and 9 months Doubly-Labeled water (DLW) are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | In-Person Caloric Restriction Arm | Remote Caloric Restriction Arm
Number analyzed (Participants) | 19 | 30
Participants | 7 | 12

2. Primary Outcome: Ability to Maintain Time Restricted Eating (TRE) Intervention
Description: This will measure the sustainability in a 9 month period of time and will be reported as the percentage of day eating within <= 8.5 hour window which is pre-specified for each participant.
Time Frame: Month 9
Measure: Median (Inter-Quartile Range); unit: % of days
Groups:
- Time Restricted Eating: Time Restricted Eating
Arm/Group | Time Restricted Eating
Number analyzed (Participants) | 34
% of days | 83.5 [68.4 to 94.6]

3. Primary Outcome: Number of Participants Who Were Retained
Description: Retention > 85%
Time Frame: Month 9
Measure: Number; unit: participants
Arm/Group | In-Person Caloric Restriction Arm | Remote Caloric Restriction Arm | Time-Restricted Eating Arm
Number analyzed (Participants) | 22 | 34 | 34
participants | 20 | 34 | 29

4. Secondary Outcome: Body Weight Change
Description: Assessed using home scales.
Time Frame: From Baseline to Month 6, and From Baseline to 9 Months
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | In-Person Caloric Restriction Arm | Remote Caloric Restriction Arm | Time-Restricted Eating Arm
Number analyzed (Participants) | 22 | 34 | 34
kg
  Change in Body Weight at 6 months | -4.47 (6.44) [-6.60 to -2.34] | -6.09 (5.58) [-7.76 to -4.41] | -1.35 (4.37) [-3.13 to 0.43]
  Change in Body Weight at 9 months | -4.44 [-6.76 to -2.10] | -6.66 [-8.49 to -4.83] | -0.94 [-2.89 to 1.02]

5. Secondary Outcome: Changes in Fat Mass
Description: Assessed by (Dual-Energy X-Ray Absorptiometry) DXA.
Time Frame: From Baseline to Month 9
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | In-Person Caloric Restriction Arm | Remote Caloric Restriction Arm | Time-Restricted Eating Arm
Number analyzed (Participants) | 22 | 34 | 34
kg | -2.92 (2.79) [-4.73 to -1.11] | -4.46 (2.46) [-5.85 to -3.07] | 0.02 (1.53) [-1.48 to 1.53]

6. Secondary Outcome: Changes in Lean Body Mass
Description: As assessed by DXA for the total lean body mass.
Time Frame: From Baseline to Month 9
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | In-Person Caloric Restriction Arm | Remote Caloric Restriction Arm | Time-Restricted Eating Arm
Number analyzed (Participants) | 22 | 34 | 34
kg | -1.73 (1.47) [-2.51 to -0.94] | -2.21 (2.03) [-2.82 to -1.60] | -0.59 (1.63) [-1.26 to 0.07]

7. Secondary Outcome: Change in Bone Mineral Density
Description: As assessed by DXA using the Hip BMD
Time Frame: From Baseline to Month 9
Measure: Least Squares Mean (95% Confidence Interval); unit: g/cm2
Arm/Group | In-Person Caloric Restriction Arm | Remote Caloric Restriction Arm | Time-Restricted Eating Arm
Number analyzed (Participants) | 22 | 34 | 34
g/cm2 | -0.01 (0.02) [-0.02 to 0.00] | -0.01 (0.03) [-0.02 to -0.00] | -0.00 (0.02) [-0.01 to 0.01]

8. Secondary Outcome: Change in Resting Energy Expenditure
Description: As assessed by Indirect Calorimetry between baseline and 9 months follow-up
Time Frame: From Baseline to Month 9
Measure: Mean (Standard Deviation); unit: Kcal
Arm/Group | In-Person Caloric Restriction Arm | Remote Caloric Restriction Arm | Time-Restricted Eating Arm
Number analyzed (Participants) | 20 | 33 | 29
Kcal | -35.3 (221.4) | -74.1 (217.3) | -94.8 (182.8)

9. Secondary Outcome: Change in Physical Activity Energy Expenditure
Description: Assessed by ActivPAL
Time Frame: From Baseline to Month 9
Measure: Mean (Standard Deviation); unit: kcals per day
Arm/Group | In-Person Caloric Restriction Arm | Remote Caloric Restriction Arm | Time-Restricted Eating Arm
Number analyzed (Participants) | 22 | 34 | 34
kcals per day | 0.42 (1.26) | 0.68 (1.19) | 0.29 (0.59)

10. Secondary Outcome: Change in Energy Intake
Description: Using doubly-labeled water (DLW). Energy intake will be calculated from Total Energy Expenditure (TEE) assessed by DLW and change in body energy stores (measured by body weight and/or DXA) according to the equation: Energy Intake = TEE + Change in body energy stores
Time Frame: From Baseline to Month 9
Measure: Mean (Standard Deviation); unit: kcals per day
Arm/Group | In-Person Caloric Restriction Arm | Remote Caloric Restriction Arm | Time-Restricted Eating Arm
Number analyzed (Participants) | 22 | 34 | 34
kcals per day | -129.5 (237.3) | -133.6 (228.7) | -45.6 (171.8)

11. Secondary Outcome: Change in Total Muscle Mass
Description: The D3-Creatine (D3Cr) method used to assess total muscle mass is completed after the participant ingests a known amount of D3-creatine (creatine with deuterium atoms replacing hydrogens) and the labeled creatine is distributed throughout the body, with approximately 98% ending up in skeletal muscle. By measuring the ratio of labeled (D3-creatinine) to unlabeled creatinine in a urine sample the total body creatine pool can be determined and total muscle mass can be calculated.
Time Frame: From Baseline to Month 9
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | In-Person Caloric Restriction Arm | Remote Caloric Restriction Arm | Time-Restricted Eating Arm
Number analyzed (Participants) | 22 | 34 | 34
kg | -1.46 [-3.51 to 0.59] | 0.64 [-0.92 to 2.20] | 1.88 [0.10 to 3.67]

12. Secondary Outcome: Change in Self-Reported Energy Intake
Description: Data will be collected and nutrients and food groups analyzed using the publicly available National Cancer Institute's Automated Self-Administered 24-Hour (ASA24) dietary assessment tool.
Time Frame: From Baseline to Month 9
Measure: Least Squares Mean (95% Confidence Interval); unit: kcals/day
Arm/Group | In-Person Caloric Restriction Arm | Remote Caloric Restriction Arm | Time-Restricted Eating Arm
Number analyzed (Participants) | 22 | 34 | 34
kcals/day | -371.4 [-612.2 to -130.6] | -244.1 [-433.0 to -55.3] | -255.6 [-452.9 to -58.3]

13. Secondary Outcome: Physical Function--Change in Walk Time
Description: 400m walk - assessed in number of seconds (unlimited time)
Time Frame: From Baseline to Month 9
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | In-Person Caloric Restriction Arm | Remote Caloric Restriction Arm | Time-Restricted Eating Arm
Number analyzed (Participants) | 22 | 34 | 34
seconds | -7.05 (40.23) [-20.02 to 5.92] | -19.76 (26.81) [-29.28 to -10.25] | -19.18 (17.58) [-29.80 to -8.56]

14. Secondary Outcome: Physical Function--Change in Grip Strength
Description: measured in kg (0-90kg)
Time Frame: From Baseline to Month 9
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | In-Person Caloric Restriction Arm | Remote Caloric Restriction Arm | Time-Restricted Eating Arm
Number analyzed (Participants) | 22 | 34 | 34
kg | -1.47 (4.34) | -0.48 (4.67) | -0.38 (5.65)

15. Secondary Outcome: Physical Function--Change in eSPPB
Description: Change in overall physical performance with total score ranging from 0 to 4 with a higher score denoting better physical function.
Time Frame: From Baseline to Month 9
Measure: Mean (Standard Deviation); unit: score
Arm/Group | In-Person Caloric Restriction Arm | Remote Caloric Restriction Arm | Time-Restricted Eating Arm
Number analyzed (Participants) | 22 | 34 | 34
score | -0.10 (0.34) | 0.08 (0.26) | -0.00 (0.22)

16. Secondary Outcome: Change in Cognitive Function--MoCA
Description: Total score ranges from 0-30 with a higher score denoting better cognitive function.
Time Frame: From baseline to Month 9
Measure: Mean (Standard Deviation); unit: score
Arm/Group | In-Person Caloric Restriction Arm | Remote Caloric Restriction Arm | Time-Restricted Eating Arm
Number analyzed (Participants) | 22 | 34 | 34
score | 1.20 (2.28) | 0.68 (2.42) | 1.17 (2.07)

17. Secondary Outcome: Change in Age-Related Biomarkers--Fasting Insulin
Description: Fasting insulin, an age-related biomarker
Time Frame: From Baseline to 9 Months
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | In-Person Caloric Restriction Arm | Remote Caloric Restriction Arm | Time-Restricted Eating Arm
Number analyzed (Participants) | 22 | 34 | 34
pmol/L | -5.60 (23.97) | -12.41 (19.91) | -2.06 (24.26)

18. Secondary Outcome: Change in Age-Related Biomarkers--interleukin-6 (IL-6)
Description: Interleukin-6 (IL-6) is an Age-related biomarker, cytokine, and key mediator of inflammation
Time Frame: From Baseline to 9 Months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | In-Person Caloric Restriction Arm | Remote Caloric Restriction Arm | Time-Restricted Eating Arm
Number analyzed (Participants) | 22 | 34 | 34
pg/mL | 1.20 (3.84) | -0.22 (1.79) | 0.30 (2.12)

19. Secondary Outcome: Change in Age-Related Biomarkers--tumor Necrosis Factor Soluble Receptor I (TNFRI)
Description: Tumor Necrosis Factor Receptor 1 (TNRFI), an Age-Related Biomarker, is a protein that acts as a receptor for TNF-alpha, a cytokin involved in inflammation.
Time Frame: From Baseline to 9 Months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | In-Person Caloric Restriction Arm | Remote Caloric Restriction Arm | Time-Restricted Eating Arm
Number analyzed (Participants) | 22 | 34 | 34
pg/mL | -3.80 (204.73) | -55.12 (281.33) | -15.52 (151.12)

20. Secondary Outcome: Change in Age-Related Biomarkers--cystatin C
Description: Change in cystatin C - An Age-Related Biomarker used to assess kidney function
Time Frame: From Baseline to 9 Months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | In-Person Caloric Restriction Arm | Remote Caloric Restriction Arm | Time-Restricted Eating Arm
Number analyzed (Participants) | 22 | 34 | 34
mg/L | -0.10 (0.21) | -0.04 (0.14) | -0.24 (1.12)

21. Secondary Outcome: Change in Age-Related Biomarkers-- CRP From Serum
Description: Change in C-reactive Protein, an Age-Related Biomarker that is used to detect inflammation in the body
Time Frame: From Baseline to 9 Months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | In-Person Caloric Restriction Arm | Remote Caloric Restriction Arm | Time-Restricted Eating Arm
Number analyzed (Participants) | 22 | 34 | 34
mg/L | 1.12 (4.47) | 0.60 (4.95) | 1.20 (6.26)

ADVERSE EVENTS:
Time Frame: AEs were collected between consent/screening and ended at study completion (approximately 9 months following start of intervention).
Arm/Group | In-Person Caloric Restriction Arm | Remote Caloric Restriction Arm | Time-Restricted Eating Arm
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 1/22 | 2/34 | 2/34
Other Adverse Events (participants affected / at risk) | 20/22 | 31/34 | 29/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In-Person Caloric Restriction Arm (N=22) | Remote Caloric Restriction Arm (N=34) | Time-Restricted Eating Arm (N=34)
Cardiac disorders - Other (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures - Other (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In-Person Caloric Restriction Arm (N=22) | Remote Caloric Restriction Arm (N=34) | Time-Restricted Eating Arm (N=34)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 3 (3) | 2 (2)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gum infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Shingles (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 2 (3) | 4 (4) | 0 (0)
Upper respiratory infection (Infections and infestations) | 6 (7) | 11 (12) | 8 (8)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 4 (5)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures - Other (Surgical and medical procedures) | 4 (4) | 2 (3) | 4 (5)
Vascular disorders - Other (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (2)
Eye disorders - Other (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (4) | 8 (11) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 7 (9) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (4) | 8 (8) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
Fatigue (General disorders) | 6 (8) | 11 (13) | 8 (10)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gum infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 3 (3) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (4) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 3 (6) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 8 (11) | 7 (8)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (7) | 18 (31) | 9 (9)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 3 (4) | 1 (1) | 2 (5)
Headache (Nervous system disorders) | 3 (3) | 4 (5) | 9 (9)
Nervous system disorders - other (Nervous system disorders) | 1 (1) | 3 (3) | 3 (3)
Presyncope (Nervous system disorders) | 4 (6) | 3 (3) | 3 (5)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2)
Depression (Psychiatric disorders) | 2 (2) | 1 (1) | 3 (3)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (2) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Surgical and medical procedures - Other (Surgical and medical procedures) | 0 (0) | 2 (2) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/42/NCT05424042/Prot_SAP_001.pdf
  • Informed Consent Form (2024-06-04): https://cdn.clinicaltrials.gov/large-docs/42/NCT05424042/ICF_000.pdf